CLINICAL TRIAL: NCT01504932
Title: Pilot Long-Term Oral Dose of Freeze-Dried Black Raspberries in Post-Surgical Appalachian Oral Cancer
Brief Title: Freeze-Dried Black Raspberries in Preventing Oral Cancer Recurrence in High At-Risk Appalachian Patients Oral Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Amit Agrawal, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-06132; NCI-2011-03189 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-15; First posted 2012-01-06 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
Keywords: black raspberry; Appalachia; oral cancer; cancer recurrence
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I: BRB Lozenge (Experimental): Former oral cancer patients receive lozenges containing freeze-dried black raspberry (BRB) powder. They will take the lozenges four times each day (QID) by mouth (PO) for up to 6 months.
  Patients will be asked to complete a baseline survey documenting any family history of cancer, tobacco, alcohol, and mouthwash use, a Head and Neck Cancer Inventory Survey (HNCI), an Insomnia Severity Index (ISI) Survey, and a Brief Fatigue Inventory (BFI) Survey.
  They will receive a trial-specific logbook to record their usages.
  Intervention: Black Raspberry (BRB) Lozenge Intervention: Survey Administration Intervention: Laboratory Biomarker Analysis
  Interventions: Dietary Supplement: BRB Lozenge; Other: Survey Administration; Other: Laboratory Biomarker Analysis; Other: pharmacological study
- Arm II: Biomarker Control (Other): Former oral cancer patients will not receive lozenges containing freeze-dried black raspberry (BRB) powder.
  Patients will be asked to complete a baseline survey documenting any family history of cancer, tobacco, alcohol, and mouthwash use, a Head and Neck Cancer Inventory Survey (HNCI), an Insomnia Severity Index (ISI) Survey, and a Brief Fatigue Inventory (BFI) Survey.
  They will receive a trial-specific logbook to record their usages.
  Intervention: Survey Administration Intervention: Laboratory Biomarker Analysis
  Interventions: Other: Survey Administration; Other: Laboratory Biomarker Analysis; Other: pharmacological study

INTERVENTIONS:
Dietary Supplement: BRB Lozenge — ARM I: Patients will be instructed to begin BRB administration and continue daily for up to 6 months.
  Other Names: BRB Troche
  Arms: Arm I: BRB Lozenge
Other: Survey Administration — Patients will complete a baseline survey documenting any family history of cancer. Patients will then provide a history of tobacco, alcohol and mouthwash use, complete the Head and Neck Cancer Inventory Survey (HNCI), the Insomnia Severity Index (ISI) Survey, and the Brief Fatigue Inventory (BFI) Survey. Patients will receive a trial-specific logbook to record their usages.
  Other Names: HNCI Head and Neck Cancer Inventory; ISI Insomnia Severity Index; BFI Brief Fatigue Inventory
Other: Laboratory Biomarker Analysis — Patients will provide blood, urine, saliva, and cheek scrape samples. These biological samples will be evaluated for the presence of BRB components (as a measure of compliance) and assessed for BRB-responsive gene expression, respectively.
  Other Names: Correlative Studies; Biological Samples
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This pilot clinical trial studies freeze-dried black raspberries (BRB) in preventing oral cancer recurrence in high at-risk Appalachian patients previously treated with surgery for oral cancer. Chemoprevention is the use of drugs natural products to keep cancer from developing, progressing, or recurring. Giving freeze-dried black raspberries may prevent oral cancer from forming or returning in oral cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct an initial early phase clinical study utilizing a high ar-risk and underserved Appalachian population who are former oral cancer patients to determine the practicability of long-term daily freeze-dried black raspberry (BRB) (BRB lozenge) administration and to gain insights into the potential prevention of recurrent oral cancer by BRBs.

SECONDARY OBJECTIVES:

I. Evaluate numerous parameters (recruitment, tolerability, adherence to study guidelines, collection of biological samples, and demographics) that will be helpful in designing a future definitive, randomized, Phase II or III clinical trial structured to assess the potential effects of long-term BRB administration.

II. Evaluate the temporal modulation of BRB-responsive gene expression that favor oral cancer chemoprevention in high at-at risk normal tissues before and after BRB administration.

III. Assess the temporal modulation of BRB-responsive gene expression and biological levels of fruit components in post-surgical oral cancer patients not exposed to BRBs.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients receive freeze-dried black raspberry lozenges orally (PO) 4 times daily (QID) for up to 6 months.

ARM II: Patients do not receive freeze-dried black raspberries lozenges.

After completion of study treatment, patients in Arm I are followed for up to 5 years and patients in Arm II are followed for up to 1 year for oral cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients from any Appalachian County with previously diagnosed, biopsy-proven, surgically resected, oral squamous cell carcinoma (SCC) (stages T1 to T4), which encompasses cancers of the oral cavity including lips, buccal mucosa, teeth, floor of the mouth and gums and those of the oropharynx consisting of the base of the tongue, soft palate, tonsillar area, and the posterior pharyngeal wall will be eligible
* Patients who have followed the advice of their physician and have been definitively treated for their tumor by any method and are currently disease free will be eligible
* Patients may be enrolled as early as their first follow-up post-operative clinic visit after their most recent surgery, but no more than 36 months post-surgery
* Patients must be able to take nutrition/medications orally
* No prior history of intolerance or allergy to berry or berry-containing products

Exclusion Criteria:

* History of intolerance (including hypersensitivity or allergy) to berry or berry-containing products
* Patients who are actively receiving adjuvant therapy (radiation, chemotherapy) will be excluded until such time as they have completed treatments
* Pregnant women; although there are no known adverse effects of black raspberries upon the fetus, if patients become pregnant during period of LBR administration, then LBR will be discontinued and patient will be removed from the study
* Inability to grant informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02-23 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | Up to 5 years
  Two side tests and confidence intervals will be constructed using the exact binomial formulation.

SECONDARY OUTCOMES:
Adherence rates in patients receiving LBR | Up to 5 years
  Adherence rates for subjects on LBR will be evaluated using 95% confidence intervals based on the exact binomial formulation (margins of error will be approximately 8% based on an expected compliance rate near 75% of subjects).
LBR-responsive gene expression before, during, and after LBR administration (Arm I) | Up to 5 years
  Reverse transcriptase polymerase chain reaction (RT-PCR) data will be analyzed on the log scale using repeated measures analysis of variance (ANOVA) models and the Bonferroni correction to adjust for the multiple inference problem
LBR-responsive gene expression in patients not exposed to LBR (Arm II) | Up to 5 years
  Reverse transcriptase polymerase chain reaction (RT-PCR) data will be analyzed on the log scale using repeated measures analysis of variance (ANOVA) models and the Bonferroni correction to adjust for the multiple inference problem.
LBR responsive gene activity and time to recurrence | Up to 5 years
  RT-PCR data will be analyzed on the log scale using repeated measures ANOVA models and the Bonferroni correction to adjust for the multiple inference problem. Genes that show changes with berries will also be compared with to a control group of 30 subjects who refuse LBR treatment but agree to be included in biomarker studies and for whom baseline alcohol and smoking history will be available

CONTACTS AND LOCATIONS:
Overall Officials: Amit Agrawal, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu